CLINICAL TRIAL: NCT00445328
Title: Prospective Randomized Phase IV Open Label Comparative Study Of Dalteparin vs Unfractionated Heparin For The Prevention Of Venous Thromboembolism (VTE) In Hospitalized Acutely Ill Medical Patients.
Brief Title: Dalteparin vs Unfractionated Heparin For The Prevention Of Venous Thromboembolism (VTE) In Hospitalized Acutely Ill Medical Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A6301080
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2009-10-02 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Venous Thromboembolism
Keywords: hospitalised acutely medically ill patients; Venous Thromboembolism, Infection, Inflammatory Bowel Diseases, Heart Failure, Congestive, Sciatica
MeSH Terms: conditions — Venous Thromboembolism; Infections; Inflammatory Bowel Diseases; Heart Failure; Sciatica | interventions — Dalteparin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Active Comparator)
  Interventions: Drug: Unfractionated heparin
- A (Experimental)
  Interventions: Drug: Dalteparin (Fragmin)

INTERVENTIONS:
Drug: Dalteparin (Fragmin) — Dalteparin 5000 IU once daily subcutaneously for 6-14 days.
  Arms: A
Drug: Unfractionated heparin — Unfractionated heparin 5000 IU thrice daily subcutaneously for 6-14 days.
  Arms: B

SUMMARY:
The purpose of this study is to compare the efficacy and safety of dalteparin vs unfractionated heparin for the prevention of VTE (Venous Thromboembolism) in hospitalized acutely ill medical patients.

DETAILED DESCRIPTION:
The study was prematurely discontinued due to delay in overall study start-up and inability to meet pre-defined protocol recruitment milestones on June 30th, 2008. There were no safety concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to 18 years
* Acute medical condition with a projected hospitalization of greater than or equal to 4 days and had less than or equal to 3 days of prior immobilization for more than two thirds of the day
* Acute congestive heart failure Class III-IV per NHYA/ Acute respiratory failure not requiring mechanical ventilation or Both
* Acute infection without septic shock/ Acute episode of inflammatory bowel disease/ Acute rheumatologic disorders/ Acute lumbar pain or sciatica or vertebral compression with at least one risk factor for VTE

Exclusion Criteria:

* Contraindications to use of anticoagulants
* Active bleeding or abnormal coagulation tests
* Recent (less than 1 month) head injury, hemorrhagic stroke, cerebral tumor or intracranial aneurysm or ischemic stroke within the last month.
* Major surgical or invasive procedure within the last month resulting in ongoing convalescence
* Lumbar or spinal puncture within last 48 hours
* S creatinine levels more than 2
* On inotropic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Thrissur, Kerala
  - Pfizer Investigational Site, Indore, Madhya Pradesh
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Kolkata, West Bengal

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6301080&StudyName=Dalteparin%20vs%20Unfractionated%20Heparin%20For%20The%20Prevention%20Of%20Venous%20Thromboembolism%20%28VTE%29%20In%20Hospitalized%20Acutely%20ill%20Medical%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalteparin: 5000 IU (International Units) dalteparin in 0.2 mL (milliliters) subcutaneously once a day (Arm A)
- Unfractionated Heparin: 5000 IU unfractionated Heparin (UFH) in 5 mL subcutaneously 3 times a day (Arm B) for 6 to 14 days.
Period: Overall Study
Arm/Group | Dalteparin | Unfractionated Heparin
Started | 42 | 42
Received Treatment | 41 (1 subject discontinued after enrollment but prior to study treatment.) | 42
Completed | 39 | 36
Not Completed | 3 | 6
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Other | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dalteparin: 5000 IU dalteparin in 0.2 mL subcutaneously once a day (Arm A)
- Total: Total of all reporting groups
Arm/Group | Dalteparin | Unfractionated Heparin | Total
Number analyzed (Participants) | 41 | 42 | 83
Age Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.6) | 60.8 (10.9) | 61.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Thromboembolic Events
Description: Confirmed thromboembolic events = 'present' if any following events are present/abnormal, otherwise = 'absent': Deep vein thrombosis measured by Color Doppler ultrasonography lower limbs; pulmonary embolism by chest xray, ventilation-perfusion scan, computed tomography pulmonary angiography; Sudden Death within 24 hours of venous thromboembolism symptoms.
Time Frame: Day 21
Population: Intent to treat (ITT) set: all subjects who were randomized, received at least 1 dose of study drug and had undergone at least 1 test of primary efficacy assessment.
Measure: Number; unit: participants
Arm/Group | Dalteparin | Unfractionated Heparin
Number analyzed (Participants) | 37 | 35
participants
  Present | 0 | 0
  Absent | 37 | 35

2. Secondary Outcome: All Cause Mortality
Description: Subjects with death from any cause: end of study.
Time Frame: Day 14, Day 21 (End of Study)
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Dalteparin | Unfractionated Heparin
Number analyzed (Participants) | 37 | 37
participants | 0 | 1
Statistical Analysis 1: Comparison: Dalteparin vs Unfractionated Heparin; Test type: Superiority or Other; p = 1.0000, Chi-squared — P-value is based on chi-square test with alpha as 0.01

3. Secondary Outcome: Stroke - Ischemic or Hemorrhagic
Description: Subjects with stroke (either ischemic or hemorrhagic) based on results of CT (computed tomographic) pulmonary angiography
Time Frame: Day 21
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Dalteparin | Unfractionated Heparin
Number analyzed (Participants) | 37 | 37
participants | 0 | 0

4. Secondary Outcome: Bleeding - Major or Minor
Description: Subjects with bleeding. Bleeding classified as major if it is: intraocular, spinal/epidural, intracranial or retroperitoneal; or if hemoglobin decreased by ≥ 2 g/dl(grams/deciliter); or if transfusion of ≥ 2 Units of blood or if significant medical or surgical intervention was required; or if it results in death. All other bleeding is classified as minor.
Time Frame: Day 21
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Dalteparin | Unfractionated Heparin
Number analyzed (Participants) | 37 | 37
participants
  Major Bleeding | 0 | 1
  Minor Bleeding | 0 | 0
Statistical Analysis 1: Comparison: Dalteparin vs Unfractionated Heparin; Major Bleeding; Test type: Superiority or Other; p = 1.0000, Chi-squared

5. Secondary Outcome: Allergic Reactions (Drug-related)
Description: Subjects with drug-related allergic reactions
Time Frame: Day 21
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Dalteparin | Unfractionated Heparin
Number analyzed (Participants) | 37 | 37
participants | 0 | 0

6. Primary Outcome: Composite of Objectively Verified Thromboembolic Events
Description: Subjects with objectively verified thromboembolic events: symptomatic proximal and distal deep vein thrombosis [DVT], asymptomatic proximal DVT, fatal or symptomatic non-fatal pulmonary embolism [PE] or sudden death within 24 hours of onset of venous thromboembolism (VTE) symptoms. Occurrence of any ='Present', otherwise = 'Absent'.
Time Frame: Day 21
Population: Intent to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Dalteparin | Unfractionated Heparin
Number analyzed (Participants) | 37 | 35
participants
  Symptomatic DVT Present | 0 | 0
  Symptomatic DVT Absent | 37 | 35
  Symptomatic Proximal DVT Present | 0 | 0
  Symptomatic Proximal DVT Absent | 37 | 35
  Symptomatic Distal DVT Present | 0 | 0
  Symptomatic Distal DVT Absent | 37 | 35
  Asymptomatic Proximal DVT Present | 0 | 0
  Asymptomatic Proximal DVT Absent | 37 | 35
  Fatal pulmonary embolism Present | 0 | 0
  Fatal pulmonary embolism Absent | 37 | 35
  Symptomatic non-fatal pulmonary embolism Present | 0 | 0
  Symptomatic non-fatal pulmonary embolism Absent | 37 | 35
  Sudden Death within 24 hours of VTE Present | 0 | 0
  Sudden Death within 24 hours of VTE Absent | 37 | 35

7. Secondary Outcome: Thrombocytopenia
Description: Subjects with thrombocytopenia (low platelets).
Time Frame: Day 21
Population: Intent to Treat (ITT)
Measure: Number; unit: participants
Arm/Group | Dalteparin | Unfractionated Heparin
Number analyzed (Participants) | 37 | 37
participants | 35 | 31
Statistical Analysis 1: Comparison: Dalteparin vs Unfractionated Heparin; Test type: Superiority or Other; p = 0.1355, Chi-squared

ADVERSE EVENTS:
Arm/Group | Dalteparin | Unfractionated Heparin
Serious Adverse Events (participants affected / at risk) | 2 | 4
Other Adverse Events (participants affected / at risk) | 7 | 7
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Dalteparin | Unfractionated Heparin
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/41 | 2/42
Chest pain (General disorders) | 0/41 | 1/42
Injection site rash (General disorders) | 0/41 | 1/42
Lobar pneumonia (Infections and infestations) | 1/41 | 0/42
Drug eruption (Skin and subcutaneous tissue disorders) | 0/41 | 1/42
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0/41 | 1/42
Diarrhoea (Gastrointestinal disorders) | 1/41 | 0/42
OTHER ADVERSE EVENTS (reported when occurring in more than 4.8% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Dalteparin | Unfractionated Heparin
Constipation (Gastrointestinal disorders) | 0/41 | 2/42
Vomiting (Gastrointestinal disorders) | 0/41 | 2/42
Pyrexia (General disorders) | 4/41 | 2/42
Blood pressure increased (Investigations) | 2/41 | 1/42
Haemoglobin decreased (Investigations) | 2/41 | 1/42
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/41 | 2/42

LIMITATIONS AND CAVEATS:
Study terminated prematurely due to delay in overall study start-up and inability to meet predefined protocol recruitment milestones; sample size too small to permit meaningful statistical analyses. No statistical analyses for all but 2 endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.